CLINICAL TRIAL: NCT07334743
Title: Identifying Biomarkers in ALS Patients Using Neuronal Derived Extracellular Vesicles
Acronym: BALNEV
Status: Recruiting | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AGN_2024_9
Record Dates: First submitted 2025-12-31; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis; ENGRAILED1
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Identification by RNA-seq of biomarkers carried by neuron-derived extracellular vesicles (NVEC) present in the blood of ALS patients, compared with NVEC from healthy controls
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with ALS
- controls without ALS

SUMMARY:
Rationale. ENGRAILED1 (EN1) is under consideration as a therapeutic approach for amyotrophic lateral sclerosis (ALS). To assess EN1 target engagement in patients, we aim to identify EN1-responsive biomarkers suitable as Prentice-style surrogate endpoints. We will discover candidates by RNA-seq of neuron-derived extracellular vesicles (NVEC) immuno-isolated from blood. Establishing such biomarkers would enable and de-risk early-phase (I/II) EN1 trials.

Primary endpoint. Discovery: RNA-seq identification of circulating NVEC-borne biomarkers that differ between sporadic ALS patients and healthy controls.

EN1 modulation: Demonstration that these biomarkers are modulated by EN1 in En1+/- mouse models and in ALS patient iPSC-derived motor neurons.

Design. Prospective cohort, N=60 (30 sporadic ALS; 30 healthy controls matched on age/sex).

Population. Adults undergoing diagnostic work-up for suspected sporadic ALS; healthy volunteers without neurological disease.

Key procedures and timeline. Baseline (M0, inpatient): ALSFRS-R, MRC, hand dynamometry, eye-movement recording (MOC); NCS/EMG (NUMIX), TMS/MEP with cortical excitability; neuropsychology; brain & spinal MRI; pulmonary function testing; CSF (10 mL) and blood (15 mL) for clinical labs and research (NVEC immunocapture → RNA-seq; proteomics).

Follow-up: M6 clinic visit (repeat clinical/electrophysiology/neuropsychology/PFTs as per care) with blood (15 mL); additional routine follow-ups at M12, M18, M24 (clinical; MOC at M12 and M24).

Controls: single visit with blood (3×5 mL EDTA) and cortical excitability; brain MRI for targeting.

Sample size. 60 participants total (30 ALS, 30 controls).

ELIGIBILITY:
Inclusion Criteria:

For patients :

Age ≥ 18 years. Diagnostic suspicion of amyotrophic lateral sclerosis (ALS). Planned inpatient admission in the HFAR neurology department for the standard diagnostic work-up as part of routine care: clinical evaluation, neuropsychological assessment, nerve conduction studies/EMG, motor evoked potentials (TMS/MEP), brain and spinal MRI, pulmonary function testing, lumbar puncture, and standard blood tests.

Explicit written informed consent to participate in the study. Affiliation with or beneficiary of a social security system.

Non-inclusion criteria:

Patient under legal protection/guardianship. Pregnant or breastfeeding woman. Active infection within the 4 weeks preceding biological sampling. Ongoing diagnosis and management of cancer.

Secondary exclusion criterion:

ALS diagnosis not confirmed.

For Healthy Controls :

Age ≥ 18 years. Explicit written informed consent to participate in the study. Affiliation with or beneficiary of a social security system.

Exclusion Criteria:

* Patient under legal protection/guardianship.
* Pregnant or breastfeeding woman.
* Diagnosed neurological disease.
* Self-reported cognitive impairment.
* Active infection within the 4 weeks prior to biological sampling.
* Current diagnosis and management of cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study Population Description. Prospective cohort of 60 adults: 30 patients undergoing inpatient diagnostic work-up for suspected sporadic ALS at the HFAR neurology department and 30 age/sex-matched healthy controls.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2029-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Identification by RNA-seq of biomarkers carried by neuron-derived extracellular vesicles (NVEC) present in the blood of ALS patients | at inclusion visit, month 6
  Identification by RNA-seq of biomarkers carried by neuron-derived extracellular vesicles (NVEC) present in the blood of ALS patients

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Fondation Adolphe de Rothschild, Paris, France